CLINICAL TRIAL: NCT00004578
Title: Phase I/II Study of ABT-378/Ritonavir in Combination With Reverse Transcriptase Inhibitors in Antiretroviral Naive HIV-Infected Patients
Brief Title: ABT-378/Ritonavir in Combination With Reverse Transcriptase Inhibitors in Antiretroviral Naïve HIV-Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: George Hanna, MD, Anti-viral Global Project Head, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 285A; M97-720
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination; Lamivudine; Stavudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Group 1, n=32 initiated with ABT-378 & ritonavir; after 3 wks stavudine and lamivudine was added.
  Interventions: Drug: Lopinavir/Ritonavir; Drug: Lamivudine; Drug: Stavudine
- 2 (Active Comparator): Group II patients (n=68) to be randomized after all Group I patients are enrolled and safety analysis is completed.
  Interventions: Drug: Lopinavir/Ritonavir; Drug: Lamivudine; Drug: Stavudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir — Lopinavir, range from 200 mg to 400 mg, every 12 hrs and Ritonavir, range from 100 mg to 200 mg, every 12 hrs
  Other Names: ABT-387; Kaletra
Drug: Lamivudine — 150 mg, every 12 hours
Drug: Stavudine — 40 mg every 12 hours

SUMMARY:
To assess the safety, tolerability and antiviral activity of lopinavir/ritonavir when administered orally in antiretroviral-HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 positive
* antiretroviral-adult males
* non-pregnant
* non-lactating females at least 18-years old with plasma HIV-1 RNA > 5000 copies/mL, who were not acutely ill

Exclusion Criteria

* History of:

  * prior antiretroviral therapy
  * significant drug hypersensitivity
  * psychiatric illness that precludes compliance
  * an active substance abuser
  * positive test results for drug abuse
  * abnormal lab test results (hemoglobin, absolute neutrophil count, platelet count, SGPT/AST or SGPT/ALT, creatinine, fasting triglycerides, significant abnormal ECG results
  * pregnancy or lactating female
  * received another investigational drug within 28 days of study initiation
  * unlikely to comply or unsuitable candidate in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1997-11; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with viral load below the limit of quantitation | 24 weeks
Time to loss of virologic response | 48 weeks

SECONDARY OUTCOMES:
Proportion of subjects with viral load below the limit of quantitation at each visit | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, MD, Study Director — Abbott
Locations (10):
- United States (10):
  - Pacific Oaks Research, Beverly Hills, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cornell Clinical Trials Unit - Chelsea Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Murphy R, King M, Brun S, Orth K, Hicks C, Eron J, Thommes J, Gulick R, Thompson M, White C, Benson C, Hammer S, Kessler H, Bertz R, Hsu A, Kempf D, Sun E, Japour A. ABT-378/ritonavir therapy in antiretroviral-naive HIV-I infected patients for 24 weeks. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:69 (abstract no 15)
- [Background] Murphy RL, Brun S, Hicks C, Eron JJ, Gulick R, King M, White AC Jr, Benson C, Thompson M, Kessler HA, Hammer S, Bertz R, Hsu A, Japour A, Sun E. ABT-378/ritonavir plus stavudine and lamivudine for the treatment of antiretroviral-naive adults with HIV-1 infection: 48-week results. AIDS. 2001 Jan 5;15(1):F1-9. doi: 10.1097/00002030-200101050-00002. PMID 11192874